CLINICAL TRIAL: NCT04202432
Title: PP3D - Prospective Combined Validation of an Algorithm for Measurement of Mean Systemic Filling Pressure and Comparison of Invasively Measured Cardiac Output Versus Cardiac Output Calculated by 3D TOE and Carotid Ultrasound.
Brief Title: Clinical Validation of Algorithms for Mean Systemic Filling Pressure and Automated Cardiac Output
Acronym: PP3D
Status: Completed | Type: Observational
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Responsible Party: Principal Investigator, L.P.B. Meijs, Cardiologist, fellow intensive care medicine, PhD candidate Intensive Care Medicine, Catharina Ziekenhuis Eindhoven
Other Study IDs: NL67389.100.18
Record Dates: First submitted 2019-12-16; First posted 2019-12-17 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Shock, Cardiogenic; Shock Hypovolemic; Hypovolemia; Cardiac Failure
Keywords: Mean Systemic Filling Pressure; Pms; Pmsf; Hypovolemia; Cardiac Output; Transpulmonary thermodilution; Transesophageal echocardiography; Volume state; Critical Care; Cardiosurgery; Intensive Care; Carotid ultrasound; Pulsed Wave; Inspiratory breath hold
MeSH Terms: conditions — Shock, Cardiogenic; Shock; Hypovolemia; Heart Failure; Premenstrual Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Coronary Artery Bypass Surgery patients: Patients undergoing coronary artery bypass surgery (on-pump / off-pump) measured perioperatively and postoperatively.
  Interventions: Diagnostic Test: Mean systemic filling pressure

INTERVENTIONS:
Diagnostic Test: Mean systemic filling pressure — Peri- and postoperative measurement of continuous cardiac output with thermodilution derived pulse contour calculated device (PiCCO).
  Estimation of mean systemic filling pressure using a computerized algorithm and by creating venous return curves with inspiratory hold maneuvers, thereby extrapolating the VR-curve until mean systemic filling pressure is calculated.
  Other Names: Measurement of cardiac output

SUMMARY:
Prospective combined clinical validation of an algorithmic calculated mean systemic filling pressure (Pms-Nav) with the gold standard for Pms (Pms calculated from venous return curves during inspiratory hold procedures with incremental airway pressures; Pms-Insp). Secondary correlation between invasive cardiac output measurement versus 3D TOE and carotid echo doppler measured cardiac output.

DETAILED DESCRIPTION:
Background of the study:

Volume-state in critically ill patients is a difficult parameter to determine, and knowledge about it could make the difference between life or death concerning proper treatment. Determination of volume state starts with adequate 3D transesophageal echocardiography (TOE) in the operation room, including with non-invasive doppler carotid artery measures. TOE is a standardly used method in cardiac surgery. Because echocardiography only gives information about volume status at a certain timepoint, a real-time continuous value reflecting volume-status is needed. "Mean systemic filling pressure (Pms)" appears to be a promising value reflecting volume status. There is a reliable, but cumbersome method available which to date serves as a gold standard to determine Pms (Pms calculated by constructing venous return curves during incremental levels of airway pressure, thereby simulating a decrease in preload --> Pms-Insp). However, this method cannot be used in daily clinical practice because it is laborious and cumbersome. Therefore there is a need for a non-invasive methods measuring Pms, which could now be determined by a computerized algorithm with the Navigator-device (Pms-Nav). It is key to compare this Pms-Nav with its gold standard (Pms-Insp) in order to establish a clinical validation for Pms-Nav.

Objective of the study:

1. Is there a good correlation between Pms-Nav and Pms-Insp?
2. Is there a good correlation between invasive continuous cardiac output measurement (by thermodilution and pulse-contour analyse detected by the PiCCO-device) and 3D transoesophageal echocardiography (TOE) and carotid echo doppler?

ELIGIBILITY:
Inclusion Criteria:

* Good left and right ventricular ejection fraction
* No significant valvular insufficiencies/stenoses
* No significant comorbidity
* Signed informed consent
* Elective coronary artery bypass surgery
* Postoperative mechanically ventilated admitted to the PACU

Exclusion Criteria:

* Withdrawal informed consent
* History of pneumonectomy of lobectomy
* Mechanical support of circulation
* COPD Gold 3 or 4
* Complications during surgery
* Postoperative bleeding >50mL/15 minutes after admission to PACU - No thoracic drain in pleura
* Postoperative pneumothorax
* Participation in other research studies/trials
* Elevated intra-abdominal surgery (>12 mmHg)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing coronary artery bypass grafting with a good left and right ventricular ejection fraction, no significant valvular insufficiencies/stenoses and no significant comorbidity.
Sampling Method: Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2019-06-24 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Clinical validation of Pms-algorithm | Hours
  To determine a correlation between Pms calculated by a computerized algorithm by Navigator(TM) (Pms-Nav) and the gold standard for determining Pms: Pms-Insp. The latter is calculated by performing inspiratory breath holds during incremental airway pressure levels thereby simulating a decrease in preload which, by extrapolating a venous return curve, leads to the true Pms when the curve intersects the x-axis (Pms-Insp).

SECONDARY OUTCOMES:
Correlation invasive continuous cardiac output and 3D-TOE / carotid artery pulsed wave CO measurement. | Hours
  Correlation between invasively measured continuous cardiac output (CO) and CO measured by a automated 3D-TOE algorithm and carotid artery PW-measured CO.

CONTACTS AND LOCATIONS:
Overall Officials: LPB Meijs, MD, Principal Investigator — Catharina Ziekenhuis Eindhoven
Locations (1):
- Catharina Hospital, Eindhoven, North Brabant, Netherlands

IPD SHARING:
Plan to Share IPD: No
No sharing

REFERENCES:
- [Derived] Meijs LPB, van Houte J, Conjaerts BCM, Bindels AJGH, Bouwman A, Houterman S, Bakker J. Clinical validation of a computerized algorithm to determine mean systemic filling pressure. J Clin Monit Comput. 2022 Feb;36(1):191-198. doi: 10.1007/s10877-020-00636-2. Epub 2021 Mar 31. PMID 33791920